CLINICAL TRIAL: NCT04020003
Title: A Clinical Study on Levosimendan Improvement of Prognosis of ARDS Patients by Optimizing Pulmonary Hemodynamics
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shenzhen Second People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20193357016
Record Dates: First submitted 2019-07-02; First posted 2019-07-15 (Actual); Last update posted 2019-07-15 (Actual); Status verified 2019-07

CONDITIONS: ARDS, Human
Keywords: Levosimendan
MeSH Terms: conditions — Respiratory Distress Syndrome | interventions — Simendan

STUDY DESIGN:
Intervention Model Description: Levosimendan group: on the basis of routine group treatment, 12.5 mg of levosimendan 5% s50ml was given on the same day, and the micro-pump was continuously pumped for 24 hours. The initial dose was 0.5 ml/ h, and if the blood pressure was not significantly decreased, the blood pressure was gradually increased to 2.4 ml/ h at the maximum dose, until the pump was over.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Routine treatment (Other): Routine treatment group: control infection, remove or control the primary disease; mechanical ventilation with low tidal volume and high PEEP mechanical ventilation strategy; strictly control volume, strengthen airway management, timely nutritional support and severe rehabilitation treatment.
  Interventions: Drug: Levosimendan

INTERVENTIONS:
Drug: Levosimendan — General treatment group: control the infection, remove or control the original disease, mechanical ventilation, small tidal volume, high PEEP mechanical ventilation strategy, strictly control the capacity, strengthen the airway management, timely nutrition support and intensive rehabilitation treatment. Levosimendan group: on the basis of routine group treatment, 12.5 mg of levosimendan 5% GS 50ml was given on the same day, and the micro-pump was continuously pumped for 24 hours. The initial dose was 0.5 ml/ h, and if the blood pressure was not significantly decreased, the blood pressure was gradually increased to 2.4 ml/ h at the maximum dose, until the pump was over. The above treatment is repeated every 7 days until the offline success or the patient leaves the ICU.

SUMMARY:
The purpose of this study was to evaluate the curative effect of Levosimendan on ARDS patients through omni-directional and multi-angle objective quantitative indexes, and to study the responsiveness of ARDS with or without right ventricular insufficiency to the treatment of Levosimendan, and to indirectly confirm whether Levosimendan had lung protective mechanism other than calcium sensitization to ARDS patients, such as inhibiting inflammatory reaction to reduce pulmonary capillary leakage and alveolar epithelial cell injury. Relaxation of bronchial smooth muscle improves pulmonary ventilation function. To provide new methods and ideas for clinical treatment of ARDS.

DETAILED DESCRIPTION:
On the basis of the above research, the investigators speculate that Levosimendan can improve cardiac function, enhance diaphragm contractility and decrease pulmonary artery through this sensitizing effect, and protect ARDS lung function by regulating the release and oxidation of inflammatory mediators and nitroso oxidative stress. The hemodynamic and pulmonary protective effects of ARDS patients were improved by regulating K-ATP channels, relieving blood vessels and bronchospasm and improving ventilation and diffusion function in ARDS patients, so as to further improve the survival rate of these patients and shorten the mechanical ventilation time and ICU stay time. The purpose of this study was to observe the effect of Levosimendan on pulmonary circulation and right ventricular function in patients with ARDS, to determine whether it can reduce the fatality rate of ARDS and shorten its ICU residence time, and to evaluate the evaluation of ARDS with or without right ventricular insufficiency and to provide a new idea and method for drug treatment of ARDS.

ELIGIBILITY:
Inclusion Criteria:

Clinical diagnosis of ARDS; joined this study with informed consents

Exclusion Criteria:

neurological and muscle diseases; Chronic severe liver and kidney failure; advanced malignant tumor; Primary left ventricular insufficiency;

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2019-07-01 (Actual); Primary Completion 2021-12-30 (Estimated); Study Completion 2022-08-30 (Estimated)

PRIMARY OUTCOMES:
APACHE II score | Admission for 24 hours
  The lowest value in the first 24 hours after entering ICU. The total score is 0~71 points. The higher the score, the more serious the disease
SOFA score | Admission for 7 days
  The total score is 0~48 points. The higher the score, the more serious the disease

SECONDARY OUTCOMES:
Mechanical ventilation time | From admission to 30 days
  how long did the patient stay in ICU
mecical expense | From admission to 30 days
  how much did the patient cost.

CONTACTS AND LOCATIONS:
Overall Officials: Feng yongwen, master, Study Chair — Shenzhen Second People's Hospital
Locations (1):
- Shenzhen Second People's Hospital, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for all primary and secondary outcome measures will be available.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Date will be available within 6 months of study completion
Access Criteria: Date assess requests will be reviewed by an external Independent Review Panel. Requestors will be required to sign a Data Access Agreement.
URL: http://www.chictr.org.cn

REFERENCES:
- [Result] Wang Q, Yokoo H, Takashina M, Sakata K, Ohashi W, Abedelzaher LA, Imaizumi T, Sakamoto T, Hattori K, Matsuda N, Hattori Y. Anti-Inflammatory Profile of Levosimendan in Cecal Ligation-Induced Septic Mice and in Lipopolysaccharide-Stimulated Macrophages. Crit Care Med. 2015 Nov;43(11):e508-20. doi: 10.1097/CCM.0000000000001269. PMID 26468714
- [Result] Gordon AC, Perkins GD, Singer M, McAuley DF, Orme RM, Santhakumaran S, Mason AJ, Cross M, Al-Beidh F, Best-Lane J, Brealey D, Nutt CL, McNamee JJ, Reschreiter H, Breen A, Liu KD, Ashby D. Levosimendan for the Prevention of Acute Organ Dysfunction in Sepsis. N Engl J Med. 2016 Oct 27;375(17):1638-1648. doi: 10.1056/NEJMoa1609409. Epub 2016 Oct 5. PMID 27705084
- Available data/document: Individual Participant Data Set: mengxinke — http://www.chictr.org.cn